CLINICAL TRIAL: NCT03796364
Title: Clinical Study of Endostatin in Improving Radiation Pneumonia and Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy director, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-008
Record Dates: First submitted 2018-12-25; First posted 2019-01-08 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Radiation Pneumonitis; Endostatin
Keywords: endostatin; Radiotherapy; Radiation pneumonitis; Radiation fibrosis
MeSH Terms: conditions — Radiation Pneumonitis; Radiation Fibrosis Syndrome | interventions — endostar protein

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): standard SRILI treatment
  Interventions: Drug: standard SRILI treatment
- observation group (Experimental): Endostar® plus standard treatment
  Interventions: Drug: Endostar; Drug: standard SRILI treatment

INTERVENTIONS:
Drug: Endostar — Patients in the observation group were treated with routine radiation pneumonia and Endostar. Endostar usage: continuous intravenous pumping of Endostar(14 doses each time) over 5 days. At week 2, 4, 6, 12, 24, 36, 52, lung functional and blood oxygen saturation was measured, chest CT and the St. George Respiratory Questionnaire (SGRQ) were assessed for quality of life at week 12, 24, 52 and before treatment; collecting the related observation indexes of patients; primary endpoint; recrudescence rate of RP; secondary endpoints; remission rate of RP and incidence rate of RF; incidence rate of RF; number of acute exacerbations and quality of life.
  Other Names: standard SRILI treatment
  Arms: observation group
Drug: standard SRILI treatment — Patients in the control group were treated with current routine radiation pneumonia. At week 2, 4, 6, 12, 24, 36, 52, lung functional and blood oxygen saturation was measured, chest CT and the St. George Respiratory Questionnaire (SGRQ) were assessed for quality of life at week 12, 24, 52 and before treatment; collecting the related observation indexes of patients; primary endpoint; recrudescence rate of RP; secondary endpoints; remission rate of RP and incidence rate of RF; incidence rate of RF; number of acute exacerbations and quality of life.

SUMMARY:
To verify the efficacy and safety of endostatin in the treatment of SRILI（symptomatic radiation-induced lung injury） and fibrosis. The results of this study are expected to be a new clinical strategy for the treatment of radiation pneumonia and fibrosis.

DETAILED DESCRIPTION:
Radiotherapy is an important treatment of lung cancer, symptomatic radiation-induced lung injury (SRILR) is the most common complications. In view of the important role of endostatin in inhibiting angiogenesis and pro-inflammatory factors, Combined with randomized controlled clinical study and small sample clinical exploration, the investigators concluded that endostatin is a new clinical technique for the treatment of radiation pneumonia（RP） and radiation fibrosis（RF）, which can reduce the recurrence rate of RP. In order to verify the efficacy and safety of endostatin in the treatment of SRILI and fibrosis, the investigators intend to use a prospective, randomized, multicenter clinical trial to classify unresectable phase III-IV Non-small cell lung cancer（NSCLC） patients with SRILI above grade 2 into the control group (standard SRILI treatment) and observation group (Endostar® plus standard treatment) on a 1:1 randomized basis. The results of this study are expected to be a new clinical strategy for the treatment of radiation pneumonia and fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients defined as NSCLC who could not be operated on, phase III-IV;
2. EOCG PS: 0-3;
3. The clinical diagnosis is RILI, with grade 2-3;
4. No major organ dysfunction, such as heart failure and chronic obstructive pneumonia;
5. No Endostar use contraindication;
6. Volunteer to participate, good compliance, can cooperate with the test observation, and sign a written informed consent.

Exclusion Criteria:

1. Patient compliance is poor and violates the test regulations;
2. Major organ dysfunction like liver and kidney occurs, such as myocardial infarction, angina pectoris, liver transaminase increased significantly;
3. Hemorrhage or thrombus occurs, anticoagulant medication is required;
4. Serious adverse drug reactions occur during treatment;
5. The patient asked to be withdrawn from the trial;
6. Other antiangiogenic drugs were used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
recrudescence rate of RP（Radiation pneumonitis） | at week12
  Patients in the observation group were treated with routine radiation pneumonia and Endostar.
  Patients in the control group were treated with current routine radiation pneumonia. Chest CT were assessed for recrudescence rate of RP at week 12. The calculation method is: number of relapse cases / total number of treatment groups × 100%; RP is classified according to CTCAE4.0, patients with grade 2 or higher are improved after treatment, and those who are assessed to be grade 2 or higher are considered recrudescence). Results are expressed as a percentage.

SECONDARY OUTCOMES:
remission rate of RP | at week 12
  Patients in the observation group were treated with routine radiation pneumonia and Endostar. Results are expressed as a percentage.
  Patients in the control group were treated with current routine radiation pneumonia. Chest CT were assessed for remission rate of RP at week 12.
incidence rate of RF（Radioactive fibrosis） | at week 12
  Patients in the observation group were treated with routine radiation pneumonia and Endostar.
  Patients in the control group were treated with current routine radiation pneumonia. Chest CT were assessed for incidence rate of RF at week 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinqiao Hospital of Chongqing, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen G, Zhu J, Jian C, Chen X, Niu K, Yang Q, Tang S, Qin S, Feng Y, Xie L, Zhuo W, Sun J. Efficacy and safety of Rh-endostatin in the treatment of radiation pneumonitis in non-small cell lung cancer. Oncologist. 2025 Nov 11;30(11):oyaf318. doi: 10.1093/oncolo/oyaf318. PMID 41014160